CLINICAL TRIAL: NCT02599311
Title: The Clinical Efficacy of Pelvic Organ Prolapse Surgery
Brief Title: the Indications and Clinical Efficacy of Pelvic Organ Prolapse Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PKUPH
Record Dates: First submitted 2015-11-01; First posted 2015-11-06 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Pelvic Organ Prolapse
Keywords: pelvic organ prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse | interventions — Tolterodine Tartrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- the efficacy (Other): transvaginal synthetic mesh
  Interventions: Device: transvaginal synthetic mesh
- the recurrence rate (No Intervention): transvaginal synthetic mesh
- the quality of life (No Intervention): transvaginal synthetic mesh
- the rate of the LUTS (Other): We use Tolterodine to improve patients' LUTS
  Interventions: Drug: Tolterodine

INTERVENTIONS:
Device: transvaginal synthetic mesh — transvaginal synthetic mesh
  Arms: the efficacy
Drug: Tolterodine — Tolterodine tartrate can improve patients' LUTS.
  Other Names: Tolterodine tartrate
  Arms: the rate of the LUTS

SUMMARY:
One thousand patients with stage>2 POP are recruited. The patients are all received surgeries,such as transvaginal synthetic mesh surgery, the sacral fixation, tissue repair surgery and colpocleisis. The patients with POP who have not undergone surgery are excluded. Postoperatively, the investigators investigate the indications and clinical efficacy of pelvic organ prolapse surgery.

DETAILED DESCRIPTION:
Postoperatively, the investigators analyze the patients' subjective and objective recurrent rates. The investigators compare the quality of life by filling out the preoperative and postoperative scoring questionnaires (PISQ 12, PFDI-20, PFIQ-7).The electrical physiological changes will be focused on. The investigators also use Overactive Bladder Symptom Score(OABss) to assess the lower urinary tract symptoms.

ELIGIBILITY:
Inclusion Criteria:

* The patients with stage>2 POP are recruited.The patients are all received surgeries, which include transvaginal synthetic mesh surgery, the sacral fixation, tissue repair surgery and colpocleisis.

Exclusion Criteria:

* The patients with POP who have not undergone surgery are excluded.

Ages: 30 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2015-08; Primary Completion 2019-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
the objective recurrent rate | one year after surgery
  The objective recurrence means postoperative stage≥2 (POP-Q) in any compartment.

SECONDARY OUTCOMES:
the rate of the lower urinary tract symptoms | one year after surgery
  We focus on lower urinary tract symptoms (LUTS), including frequent micturition, urgent urination, cough (or sneezing) leakage, dysuria, and urinary incontinence.
the quality of life questionnaires | one year after surgery
  The QOL questionnaires include PFDI-20 and PFIQ-7.

CONTACTS AND LOCATIONS:
Overall Officials: Jianliu Wang, professor, Study Chair — department of Gynecology, Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China